CLINICAL TRIAL: NCT05712096
Title: An Observational Study to Assess the Real-world Effectiveness of EVUSHELD™ (Tixagevimab/Cilgavimab) as Pre-exposure Prophylaxis Against COVID-19 Among Immunocompromised Patients in Israel
Brief Title: eVusheld Assessment reaL wORld Effectiveness in Israel Clalit Health Services
Acronym: VALOR C19 IL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: D8850R00002
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: SARS-CoV-2; COVID-19
Keywords: SARS-CoV-2; COVID-19; Immunocompromised Patients; Pre-exposure Prophylaxis Against COVID-19; Evusheld
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- EVUSHELD Arm: Individuals given EVUSHELD for pre-exposure prophylaxis
  Interventions: Drug: EVUSHELD
- Concurrent Control Arm: Individuals eligible for EVUSHELD pre-exposure prophylaxis but did not receive Evusheld

INTERVENTIONS:
Drug: EVUSHELD — EVUSHELD (AZD 7442, Tixagévimab/Cilgavimab)
  Groups: EVUSHELD Arm

SUMMARY:
An AstraZeneca-sponsored observational, electronic healthcare record (EHR)-embedded retrospective cohort study to assess the real-world effectiveness of EVUSHELD against SARS-CoV-2 infection, COVID-19-related hospitalization, and other COVID-19 related outcomes in the total EVUSHELD eligible patient population in the Clalit Health Services in Israel.

DETAILED DESCRIPTION:
This a Phase IV observational, secondary data study to assess the effectiveness of EVUSHELD in preventing COVID-19 infection and severe outcomes using the electronic medical records from the nationwide integrated health system.

The study is designed as an AstraZeneca-sponsored observational, electronic healthcare record (EHR)-embedded retrospective cohort study to assess the real-world effectiveness of EVUSHELD against SARS-CoV-2 infection, COVID-19-related hospitalization, and other COVID-19 related outcomes in the total EVUSHELD eligible patient population in the Clalit Health Services in Israel.

ELIGIBILITY:
Individuals who meet all criteria below will be included. The eligibility criteria aligns with the guidelines of the Israeli Ministry of Health

Inclusion criteria:

* Aged 12 years and older as of the date of receipt of EVUSHELD
* No record of infection or SARS-CoV- hospitalization within last 90 days prior to the index date
* Individuals who are moderate/severe immune compromised due to a medical condition or receipt of immunosuppressive medications or treatments and may mount an adequate immune response to COVID-19 vaccine:
* Hypogammaglobinemia patients regularly treated with immunoglobulins
* Patients treated with B-cell depleting therapy, including for example such anti-CD20 as rituximab, obinatuzumab, ofatumumab, veltuzumab, Y-ibritumomab tiuxetan or ocrelizumab, even without malignant disease, up to six months from treatment.
* Patients that are treated with B-cell depleting therapy (i.e. anti CD20, rituximab, Y-ibritumomab tiuxetan, veltuzumab, ofatumumab, obinatuzumab, ocrelizumab), without a malignant disease
* Bone marrow transplant (up to a year from the BMT) from outside donors, or with GVHD grades 3-4.
* Bone marrow transplant (up to a 6 months after the BMT) from self
* Patients after (CAR) T-cell therapy (chimeric antigen receptor T-cell therapy) up to 6 months from the treatment.
* Lungs transplant recipients
* Solid organ transplant recipients (who has any kind of transplant) or those who received ATG (anti thymocyte globulin) over the last 6 months
* Patients with aggressive lymphoma.
* Multiple Myeloma patients that have active disease, and on treatment at the time of study initiation.

Individuals who meet the criterion below will be excluded:

Per the current FDA EUA, individuals currently infected with SARS-CoV-2 are not eligible for EVUSHELD as PrEP. Therefore, in the main analysis, individuals who meet the following criteria will also be excluded.

Exclusion Criteria:

* With evidence of COVID 19 (i.e., a positive diagnostic test, or COVID-19 diagnosis code) in the period of 90 days before (pseudo) index date OR
* With evidence of SARS-CoV-2 infection on the (pseudo) index date or anytime within the 6-day period immediately following this date (i.e., index date to index date+6)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All EVUSHELD PrEP-eligible patient population in the Clalit Health Services system
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Hospitalisation due to COVID-19 | up to 6 months
  Any record of admission to hospital that was reported to the Israeli MOH as hospitalization due to SARS-CoV-2
All-cause mortality | up to 6 months
  All-cause deaths reported in the patient's record

SECONDARY OUTCOMES:
Documented SARS-CoV-2 Infection, COVID-19 related mortality, Severe COVID-19 | 6 months and 12 months
  SARS-CoV-2 diagnostic test (eg, PCR, nucleic acid amplification, antigen) OR medical encounter resulting in a diagnosis code for COVID-19b OR medical encounter resulting in a code for isolation due to COVID-19
COVID-19 mortality | 6 months and 12 months
  Any record indicating death due to COVID-19 or record of death certificate mentioning SARS-CoV-2 as cause of death.
COVID-19-related healthcare resource utilization (HCRU) | 6 months
  Any record of COVID-19 hospitalisation, ICU admission, mechanical ventilation and prescriptions of therapies for COVID-19
COVID-19-related healthcare resource utilization | 6 months
  Any record of hospital admission including hospital lenght of stay, ICU, mechanical ventilation, prescription/dispensations of antiviral drugs used for COVID-19 drugs
SAEs/AESIs | 6 months
  Any record of Serious Adverse Events (SAEs) or Adverse Events of Special Interests (AESIs) up to 6 months following initiation of Evusheld
Adverse events (AEs) | 12 months
  Any record of Adverse events up to 12 months following initiation of Evusheld

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850R00002&attachmentIdentifier=41cb241f-eab4-4b74-831f-d78735fb5dc6&fileName=D8850R00002-CSR_Synopsis_Redacted_final.pdf&versionIdentifier=